CLINICAL TRIAL: NCT00005468
Title: Lipid Variability--Influence of Stress
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4913; R01HL043041 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia

SUMMARY:
To investigate the variability of lipids and specifically the effects of stress on serum triglyceride levels, total cholesterol, HDL, and LDL in a 2.5 year epidemiological study.

DETAILED DESCRIPTION:
BACKGROUND:

While researchers had documented some of the behavioral contributors to fluctuation in individuals' lipid levels (e.g., nutrition patterns, smoking, exercise), little attention had been given to psychosocial stress. Early reports utilizing accountants, race car drivers, and air traffic controllers provided some uncontrolled data associating stress with cholesterol increases. Yet, no empirical research on stress that concomitantly examined other related influences was available. This paucity of data was probably due to lack of objective measures of stress and difficulty in measuring lipid subfractions.

DESIGN NARRATIVE:

Based on the results of their pilot study, and their research observations, the investigators predicted significant positive associations between stress level and triglycerides. A total of 228 public accountants (148 men and 80 women to provide comparable power between the sexes) were recruited from the greater Birmingham, Alabama area. Participants were evaluated monthly for 18 months, across three stressful and non-stressful work intervals (i.e., tax seasons). The investigators also collected data (during this same time frame) to closely monitor the following variables that affect lipids: dietary intake (including alcohol, caffeine, total calories, total fat, saturated fat, and dietary cholesterol), smoking, and physical activity, and oral contraceptive use, pregnancy status and menstrual stage among the women. Additionally, a substudy presented a unique opportunity for them to investigate the relation between stress and triglyceride-rich lipoproteins in the formation of foam cells.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-07; Study Completion 1992-12 (Actual)